CLINICAL TRIAL: NCT06861985
Title: The Effects of High-Frequency Multiband Harmonic Electromagnetic Stimulation (HFMH-EMS) on Ocular Artery Circulation After Prolonged Smartphone Usage
Brief Title: Effects of HFMH-EMS on Ocular Artery Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202304EM005
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Ocular Surface Disease; Central Retinal Artery Occlusion
MeSH Terms: conditions — Retinal Artery Occlusion

STUDY DESIGN:
Intervention Model Description: This study is a randomized double-blind controlled trial. All participants who meet the inclusion criteria are randomly assigned to either the "high-frequency multi-band harmonic electromagnetic stimulation device group" as the experimental group or the "placebo device group" as the control group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): high-frequency multi-band harmonic electromagnetic stimulation device group
  Interventions: Device: BOBY
- control group (Placebo Comparator): placebo device group
  Interventions: Other: Control

INTERVENTIONS:
Device: BOBY — high-frequency multi-band harmonic electromagnetic stimulation device
  Arms: experimental group
Other: Control — placebo group
  Arms: control group

SUMMARY:
Investigated the effects of high-frequency multi-band harmonic electromagnetic stimulation on ophthalmic and central retinal artery circulation.

DETAILED DESCRIPTION:
This study investigated the effects of prolonged smartphone usage for over 90 minutes on ophthalmic and central retinal artery circulation before and after smartphone use and compared the effects with versus without intervention by high-frequency multi-band harmonic electromagnetic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 65 years old

Exclusion Criteria:

* hypertension
* diabetes
* heart disease
* eye-related diseases

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Peak Systolic Velocity (PSV) | At the first visit and after 90 minutes usage of device.
  peak systolic velocity (PSV) of the ophthalmic artery (OA) were measured using color Doppler ultrasound of the eye arterial blood flow (EPIQ Elite ultrasound system, PHILIPS).
End Diastolic Velocity (EDV) | At the first visit and after 90 minutes usage of device.
  end diastolic velocity (EDV) of the ophthalmic artery (OA) were measured using color Doppler ultrasound of the eye arterial blood flow (EPIQ Elite ultrasound system, PHILIPS).
Central Retinal Artery (CRA) | At the first visit and after 90 minutes usage of device.
  Central Retinal Artery (CRA) were measured using color Doppler ultrasound of the eye arterial blood flow (EPIQ Elite ultrasound system, PHILIPS).

CONTACTS AND LOCATIONS:
Locations (1):
- National Central University, Hsinchu, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No